CLINICAL TRIAL: NCT05206656
Title: Safety and Efficacy of Eribullin or Eribulin Combined With Anlotinib in Metastatic Breast Cancer Patients: An Open-Labeled, Single-center, Prospective Study
Brief Title: Safety and Efficacy of Eribullin or Eribulin Combined With Anlotinib in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYS-20200305
Record Dates: First submitted 2021-12-16; First posted 2022-01-25 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eribulin mesylate (Placebo Comparator): Metastatic breast cancer patients receive eribulin mesylate injection alone. The dosage is 1.4mg/m2 for one cycle. Injection is performed on Day 1 and Day 8 of a treatment cycle. Patients receive Eribulin untill progression.
  Patients were observed for at least 6 months but no longer than 18 months.
  Interventions: Drug: Eribulin Mesylate
- Eribulin mesylate combined with Anlotinib (Experimental): Metastatic breast cancer patients receive Eribulin mesylate combined with Anlotinib. The dosage of Eribulin mesylate is 1.4mg/m2 for one cycle. Injection is performed on Day 1 and Day 8 of a treatment cycle.
  Anlotinib dosage is 12mg per day for consecutive 14 days (21 days per cycle). Patients receive Anlotinib untill progression.
  Patients were observed for at least 6 months but no longer than 18 months.
  Interventions: Drug: Eribulin Mesylate; Drug: Anlotinib

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate injection is performed on Day 1 and Day 8 of each treatment cycle (21 days per cycle). Patients were treated for six cycles, except disease progression (PD) or treatment stop for other reasons, such as severe adverse effects.
Drug: Anlotinib — 12 mg Anlotinib is administered for continuous 14 days in 21 day cycles. Patients received Anlotinib untill disease progression.
  Arms: Eribulin mesylate combined with Anlotinib

SUMMARY:
Eribulin is the promising agent for late-line metastatic breast cancer patients. The aim of this Phase II, double-arm, open-label and prospective clinical trial is to assess the efficacy and safety of Eribullin or Eribulin combined with Anlotinib in patients with metastatic breast cancer

DETAILED DESCRIPTION:
The aim of the double-arm, open-label, phase II clinical trial is to assess efficacy and safety of Eribulin or Eribulin combined with Anlotinib in metastatic breast cancers. The investigator hypothesize that both Eribulin and Eribulin combined with Anlotinib may be an effective alternative treatment for metastatic breast cancers. In addition, Eribulin combined with Anlotinib might be able to improve the treatment response and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, voluntary consent and signed written informed consent
* ECOG 0~2
* Pathologically diagnosed HER2-negative breast cancer patients with radiologically confirmed locally advanced (stage IIIB or IIIC) or metastatic (stage IV) breast cancer; HR-positive patients were permitted
* At least one measurable disease lesion before treatment
* Never receive Eribulin Mesylate treatment or anti-angiogenetic therapies before recruitment
* Anticipated survival time is longer than three months
* Brain metastases with stable disease or without clinical symptom
* Blood routine test, liver and kidney function test meet the following criteria: PLT > 100g / L, Hb > 9g / L, Neutrophil > 2.0 g/L; AST and ALT < 2.5 upper limit of normal (ULN); Cr < 1.0 ULN; TBIL < 1.5ULN
* Previously treated with anthracycline-based and taxane-based chemotherapy regimens (at least one line of chemotherapy in the metastatic setting or the recurrence time is less than 1 year from the end of adjuvant or neoadjuvant chemotherapy); for HR-positive/HER2-negative patients, progressed after at least one line of endocrine therapy
* For women with fertility, the pregnancy test before administration was negative, and agreed to take appropriate measures to avoid pregnancy during the study treatment and at least half a year after the end of treatment; Men agreed to take appropriate contraceptive measures during the study treatment and at least half a year after the end of the treatment.

Exclusion Criteria:

* Pregnant or lactating women
* Active infection requiring systemic treatment
* HIV positive
* Suffering from or suspected of suffering from central neuromuscular system diseases
* Serious heart disease; uncontrollable hypertension; history of heavy hemorrhea；recent operation within three months
* The investigator considered that the patient was not suitable for in this study, with any other situation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | through study completion, up to 6 months.
  The time from the date of recruitment to the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | At the end of Cycle 2 (42 days).
  The total rate of CR+PR+SD after the completion of two cycles of treatment
Overall survival (OS) | through study completion, an average of 2 year
  The survival time from the date of recruitment to the date of death from any cause
Objective response rate (ORR) | At the end of Cycle 2 (42 days).
  The total rate of CR+PR after the completion of two cycles of treatment
Adverse Events | through study completion, up to 6 months.
  All adverse events [including adverse events (AE / SAE) and ADR (adverse drug reactions)] will be collected when known. The classification of adverse reactions shall refer to CTCAE5.0 in case of adverse events / reactions. In case of serious adverse events, the investigators must immediately take necessary treatment measures to protect the safety of subjects. All adverse events / reactions should be tracked and observed. If the adverse events have not recovered, the investigator shall continue to give necessary treatment, report and record, and deal with special cases according to the management opinions of relevant departments.
Patient Report Outcome (PRO) | through study completion, up to 6 months.
  HRQoL was assessed using FACT-B at baseline and months 1,3 ,6, 9 and 12 (end of treatment). Questionnaires were administered in the local language and completed independently by patients using paper document during visits to their reference center and before any clinical procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No